CLINICAL TRIAL: NCT04079777
Title: Relationship Between Acute Severe Pancreatitis and Mitochondrial DNA
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: First People's Hospital of Chenzhou (Other)
Responsible Party: Principal Investigator, Xingui Dai, Critical Care Medicine, First People's Hospital of Chenzhou
Other Study IDs: severe acute pancreatitis
Record Dates: First submitted 2019-08-30; First posted 2019-09-06 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Severe Acute Pancreatitis
Keywords: Mitochondrial DNA ;mtDNA;; Acute pancreatitis;SAP;severe acute pancreatitis;; Acute pancreatic necrosis;; Inflammatory necrosis;
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Clinical diagnosis of severe acute pancreatitis: 1, with typical clinical manifestations, such as abdominal pain or nausea and vomiting, accompanied by epigastric tenderness or peritoneal irritation.
  2. Pancreatin content in serum, urine or abdominal cavity puncture fluid increases.
  3. Image examination (ultrasound, CT) showed pancreatic inflammation or pancreatic inflammation seen by surgery or confirmed by autopsy pathology.
  4, can except other similar clinical manifestations of lesions.
  Interventions: Drug: Clinical treatment
- mtDNA: Mitochondrial DNA is the genetic material in mitochondria. Mitochondria can produce energy (ATP) for cells, which is a special form of ribonucleic acid found in mitochondria of cells. Mitochondria are organelles that provide energy (ATP) to cells. There are usually many DNA molecules in a mitochondria.
  They carry their own DNA--mtDNA, and mutations in these genes can cause mitochondrial diseases. Although the symptoms of the disease are changeable, organs that consume more energy, such as brain, muscle and heart, are usually affected. Since mitochondria are transmitted through egg cells, related diseases will be inherited from the mother.
  Interventions: Drug: Clinical treatment

INTERVENTIONS:
Drug: Clinical treatment — Liquid Resuscitation, Anti-infection
  Other Names: Clinical treatment such as fluid infusion

SUMMARY:
Plasma mtDNA analysis aids in predicting pancreatic necrosis in severe acute pancreatitis patients.After the onset of severe acute pancreatitis, pancreatic necrosis and the content of mtDNA in plasma will increase, showing a significant positive correlation.

DETAILED DESCRIPTION:
Acute pancreatitis is an acute inflammatory disease of the pancreas characterized by the sudden onset of abdominal pain, elevated serum amylase, and edema or necrosis of the pancreas. The clinical course of AP is generally mild; however, nearly 25% of patients progress into severe AP which consists of organ failure and/or pancreatic necrosis. Although advances in the diagnosis and management have been made, AP remains a major health issue to the society. PNec is a major complication of AP which manifests as non-opacified parenchyma with intravenous contrast, as identified via contrast-enhanced CT scan. Patients with PNec are more likely to develop pancreatic infection and suffer a greater risk for mortality . Currently, CECT scans remain the "gold standard" to diagnosis PNec clinically. However, the extent of PNec is best seen about 3 days after the presentation of disease and may be missed in early CT scan. In addition, repeated CT scanning is not convenient to monitor changes in necrosis, most notably for those who are receiving mechanical ventilation or hemofiltration.The clinical diagnosis of AP is based on the presence of the following features: abdominal pain; serum amylase and/or lipase levels three times higher than the upper limit of normal; and characteristic findings of AP on CT scan.

Specific plasma biomarkers in predicting pancreatic necrosis (PNec) are needed in treating acute pancreatitis (AP). Aims To investigate the prognostic value of plasma mitochondrial DNA fragments (mtDNA) in patient with AP for PNec. Methods AP patients with symptoms onset within 72 h were prospectively enrolled.The conclusions elevated plasma mtDNA content in AP patients may be used as a more accurate early predictor of PNec in contrast to traditional CRP.

Normally,human mtDNA is strictly contained in mitochondria and not exposed to the innate immune system even following cell apoptosis. However, in times of cell death elicited by stress (e.g., trauma and sepsis), mtDNA is released into systemic circulation and leads to an array of inflammatory reactions. Elevated mtDNA levels have been reported in a variety of clinical situations, including trauma, severe sepsis, and cancer. As PNec is caused by intracellular activation of digestive enzymes and autodigestion, we assumed that circulating mtDNA levels could be used as a biomarker for early detection of PNec.

Research methods and steps:cell culture and mtDNA extraction、mtDNA detection、statistical analysis、results.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of severe acute pancreatitis
* Admission time less than two days

Exclusion Criteria:

* Malignant Tumor
* Positive confirmed pregnancy or urinary pregnancy test
* Acute liver failure
* Immunosuppressive state
* Hormone use
* Transplantation
* Death within seven days
* Blood transfusion over 1000ml in seven days
* Missing Visits
* Incomplete information
* Family Requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Acute severe pancreatitis patients admitted to hospital emergency department
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
mtDNA | one day after onset to clinical cure
  mtDNA content In plasma

CONTACTS AND LOCATIONS:
Overall Officials: Dixian DX, Study Director — First People's Hospital of Chenzhou
Locations (1):
- The First Hospital of Chenzhou, Chenzhou, Hunan, China